CLINICAL TRIAL: NCT02553109
Title: The Risk of Rupture or Growth in Patients With Small Unruptured Paraclinoid Aneurysm: Paraclinoid ANeurysm Prospectively Driven ObseRvational Analysis (PANDORA) Study
Brief Title: Paraclinoid ANeurysm Prospectively Driven ObseRvational Analysis (PANDORA) Study
Acronym: PANDORA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); DongGuk University (Other); Inje University (Other); Jeju National University Hospital (Other); KangWon National University Hospital (Other); Gyeongsang National University Hospital (Other); Soonchunhyang University Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Eun Kim, Professor, Seoul National University Hospital
Other Study IDs: SNUH-001
Record Dates: First submitted 2015-08-20; First posted 2015-09-17 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Unruptured Aneurysm of Carotid Artery
Keywords: small paraclinoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- small unruptured paraclinoid aneurysm: Patients with newly diagnosed, small (less than 5mm) unruptured paraclinoid aneurysms who will visit one of the study centers during the period from January 2015 to February 2017. Patients would be eligible for enrollment if they were 20 years of age or older and had an unruptured paraclinoid aneurysm that is less than 5 mm in the largest dimension. All patients who would visit a study center during the enrollment period and meet these criteria will be asked to join the study. The cohort will consists of patients who agree to participate. Target population of this study is 645 aneurysms.

SUMMARY:
The optimal consensus concerning treatment of incidental small paraclinoid unruptured intracranial aneurysms (UIAs) remains controversial. The aim of this prospective study is to reveal the natural history of small paraclinoid UIAs with the goal of informing the treatment plan.

DETAILED DESCRIPTION:
A prospective observational study will be conducted in 13 Korean centers enrolling a consecutive series of 645 patients with small paraclinoid unruptured intracranial aneurysms (UIAs) from 2015 to 2017.

The investigators defined the cohort population as adults(20 years old or more) with small (less than 5mm) unruptured paraclinoid aneurysm. To determine the growth rate and risk factors, the angiographic features based on MRA or CTA(ex) size, arterial relationship, multiplicity)and the clinical characteristics (ex) age, hypertension (HTN), diabetes mellitus(DM), Hyperlipidemia, smoking) are recorded at initial visit, 1 year, 2years, 3years, and 5years.

The cumulative risk and the risk factors of aneurysmal rupture and growth will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed small unruptured paraclinoid aneurysms who agreed to participate.
* 20years old or more
* less than 5mm in maximum diameter
* neurological status of patients should be satisfied with less than modified Rankin score 2 or more than 70 in Karnofsky performance score

Exclusion Criteria:

* patients had previous subarachnoid hemorrhage that could be related to the rupture of paraclinoid aneurysm.
* traumatic, infectious or dissecting aneurysms
* fusiform aneurysms
* aneurysms that related to other vascular disease or brain tumor
* aneurysm that associated with the atherosclerotic change of a parent artery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invastigators defined the cohort population as adults( more than 20 years old) with newly diagnosed small (less than 5mm) unruptured paraclinoid aneurysm who agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2015-01; Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of increased maximal diameter of enrolled paraclinoid aneurysms on follow up MRA or CTA | within 5years after enrollment
  If, the maximal diameter(in mm) of aneurysm which is measured by 1 neurosurgeon and 1 neuroradiologist on follow up MRA or CTA (1,2,3,5 year follow up) is 1.5 times bigger than on initial MRA or CTA, investigators will decide that the aneurysm is increased.
Number of rupture of enrolled paraclinoid aneurysms | within 5years after enrollment
  annual rupture rate

SECONDARY OUTCOMES:
Mortality rate of enrolled patients(related to rupture of aneurysm or not) | within 5years after enrollment
  death due to ruptured aneurysm
Number of participants with worsened modified Rankin scale score | within 5years after enrollment
  from 0(No symptom at all) to 6(Dead)
Number of participants with worsened Karnofsky Performance Status scale | within 5years after enrollment
  from 0(Dead) to 100(Normal)
Treatment(due to growth or rupture) rate of enrolled aneurysms | within 5years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Eun Kim, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (8):
- South Korea (8):
  - KangWon National University Hospital, Chuncheon, Gangwon-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Sungkyunkwan University Samsung Medical center, Seoul, Kangnam
  - DongGuk University, Ilsan, Kyungkido
  - Seoul National University Bundang Hospital, Seongnam-si, Kyungkido
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Soonchunhyang University Hospital - Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeon JS, Ahn JH, Huh W, Son YJ, Bang JS, Kang HS, Sohn CH, Oh CW, Kwon OK, Kim JE. A retrospective analysis on the natural history of incidental small paraclinoid unruptured aneurysm. J Neurol Neurosurg Psychiatry. 2014 Mar;85(3):289-94. doi: 10.1136/jnnp-2013-305019. Epub 2013 Jun 18. PMID 23781005
- [Background] Barami K, Hernandez VS, Diaz FG, Guthikonda M. Paraclinoid Carotid Aneurysms: Surgical Management, Complications, and Outcome Based on a New Classification Scheme. Skull Base. 2003 Feb;13(1):31-41. doi: 10.1055/s-2003-820555. PMID 15912157
- [Background] Juvela S, Poussa K, Lehto H, Porras M. Natural history of unruptured intracranial aneurysms: a long-term follow-up study. Stroke. 2013 Sep;44(9):2414-21. doi: 10.1161/STROKEAHA.113.001838. Epub 2013 Jul 18. PMID 23868274
- [Background] Sonobe M, Yamazaki T, Yonekura M, Kikuchi H. Small unruptured intracranial aneurysm verification study: SUAVe study, Japan. Stroke. 2010 Sep;41(9):1969-77. doi: 10.1161/STROKEAHA.110.585059. Epub 2010 Jul 29. PMID 20671254
- [Background] UCAS Japan Investigators; Morita A, Kirino T, Hashi K, Aoki N, Fukuhara S, Hashimoto N, Nakayama T, Sakai M, Teramoto A, Tominari S, Yoshimoto T. The natural course of unruptured cerebral aneurysms in a Japanese cohort. N Engl J Med. 2012 Jun 28;366(26):2474-82. doi: 10.1056/NEJMoa1113260. PMID 22738097
- [Background] Wiebers DO, Whisnant JP, Huston J 3rd, Meissner I, Brown RD Jr, Piepgras DG, Forbes GS, Thielen K, Nichols D, O'Fallon WM, Peacock J, Jaeger L, Kassell NF, Kongable-Beckman GL, Torner JC; International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms: natural history, clinical outcome, and risks of surgical and endovascular treatment. Lancet. 2003 Jul 12;362(9378):103-10. doi: 10.1016/s0140-6736(03)13860-3. PMID 12867109